CLINICAL TRIAL: NCT03104179
Title: Removal of Cytokines in Patients Undergoing Cardiac Surgery With CPB (The REMOTE Study)
Brief Title: Removal of Cytokines in Patients Undergoing Cardiac Surgery With CPB
Acronym: REMOTE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Klinikum Nürnberg (Other)
Collaborators: CytoSorbents, Inc (Industry)
Responsible Party: Principal Investigator, PD Dr. med. Giuseppe Santarpino, PD, Dr. med, Klinikum Nürnberg
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1_15B
Record Dates: First submitted 2015-06-16; First posted 2017-04-07 (Actual); Last update posted 2017-04-07 (Actual); Status verified 2017-03

CONDITIONS: Extracorporeal Circulation; Hemofiltration

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): CPB with Cytosorb
  Interventions: Device: Cytosorb Adsorber
- Control (No Intervention): CPB without Cytosorb (Control)

INTERVENTIONS:
Device: Cytosorb Adsorber — Cytokine adsorption during CPB
  Arms: Treatment

SUMMARY:
In a lot of cases during cardiac surgery cardiopulmonary bypass initiates SIRS due to release of cytokines during immunological response.

They are induced by different types of inductors ( intrinsic and extrinsic). High levels of inflammation markers like TNF-a, IL 6 and IL 10 as well as TGF-ß are detectable after 2 hours of surgery.

Beside the inflammation acute phase parameters like fibrinogen, ferritin are increased. These changes lead to rheology impairments.

These strong reactions lead to dysfunction of different organs possibly culminating in a multi organ failure.

There is a correlation between amounts of cytokines and mortality. Often AKI occurs after CPB with a rate of about 30%. Dysfunctions of organ function are often connected with increased mortality, prolonged mechanical ventilation , septic complications, increased catecholamine dosages and prolonged length of ICU stay.

Use of cytokine adsorption within the extracorporeal circuit during CBP can affect the circulating cytokine levels during and after CPB and lead to a diminished inflammatory response, acute phase reaction as well as reduction of organ failure.

DETAILED DESCRIPTION:
In a lot of cases during cardiac surgery cardiopulmonary bypass initiates SIRS due to release of cytokines during immunological response.

They are induced by different types of inductors ( intrinsic and extrinsic). High levels of inflammation markers like TNF-a, IL 6 and IL 10 as well as TGF-ß are detectable after 2 hours of surgery.

Beside the inflammation acute phase parameters like fibrinogen, ferritin are increased. These changes lead to rheology impairments.

These strong reactions lead to dysfunction of different organs possibly culminating in a multi organ failure.

There is a correlation between amounts of cytokines and mortality. Often AKI occurs after CPB with a rate of about 30%. Dysfunctions of organ function are often connected with increased mortality, prolonged mechanical ventilation , septic complications, increased catecholamine dosages and prolonged length of ICU stay.

Use of cytokine adsorption within the extracorporeal circuit during CBP can affect the circulating cytokine levels during and after CPB and lead to a diminished inflammatory response, acute phase reaction as well as reduction of organ failure.

Official Title: Removal of Cytokines in patients undergoing cardiac surgery with CPB ( The REMOTE Study)

Study type: Interventional Study design: randomized, controlled Endpoint Classification: Efficacy study Interventional Model: Parallel assignment Masking: Single blinding ( Subject) Primary purpose: Treatment

Patients who have an elective cardiac surgery with an expected CPB duration > 75 min ( e.g. valve surgery, CABG, combined procedures, redo) will be enrolled into the study after a giving informed consent.

Selection of patients are directed by randomization. Patient which drop out will be replaced.

ELIGIBILITY:
Inclusion Criteria:

* Elective cardiac surgery with CPB
* Signed informed consent
* CPB time > 75 min.
* Comorbidities:
* diabetes mellitus
* CHF, NYHA class 1 and 2
* liver dysfunction (1, 2)
* kidney dysfunction (1, 2)
* hypertension
* arteriosclerosis

Exclusion Criteria:

* Age < 65 years
* Declined informed consent
* Planed temperature < 32 C
* Emergency surgery
* Preexisting renal replacement therapy
* Preexisting kidney transplantation
* Administration of immunosuppressants like steroids
* AIDS with CD 4 < 200/
* Participation in other trials

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2017-05 (Estimated); Primary Completion 2019-05 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
Cytokine levels following CPB | 72 hours
  Evaluation of cytokine adsorber effect on cytokine levels intra- and post

SECONDARY OUTCOMES:
Intra- and postoperative catecholamine dosages | until ICU discharge, expected average 4 days
  Impact of intraoperative Cytokine adsorption on hemodynamic stability
postoperative renal failure necessitating RRT | until ICU discharge, expected average 4 days
  Impact of intraoperative Cytokine adsorption on postoperative organ function
Level of ferritin | 72 hours
  Impact of intraoperative Cytokine adsorption on iron metabolism
Level of transferrin | 72 hours
  Impact of intraoperative Cytokine adsorption on iron metabolism
Level of haptoglobin | 72 hours
  Impact of intraoperative Cytokine adsorption on iron metabolism
Length of ICU stay | until discharge from ICU, expected average 4 days
  Impact of intraoperative Cytokine adsorption on postoperative patient course
Length of hospital stay | up to hospital discharge, expected average 14 days
  Impact of intraoperative Cytokine adsorption on postoperative patient course

OTHER OUTCOMES:
Mortality | 28 days
  Impact of intraoperative Cytokine adsorption on postoperative patient course

CONTACTS AND LOCATIONS:
Locations (1):
- Klinikum Nürnberg - Nuremberg Hospital, Nuremberg, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Levy JH, Tanaka KA. Inflammatory response to cardiopulmonary bypass. Ann Thorac Surg. 2003 Feb;75(2):S715-20. doi: 10.1016/s0003-4975(02)04701-x. PMID 12607717
- [Background] Allan CK, Newburger JW, McGrath E, Elder J, Psoinos C, Laussen PC, del Nido PJ, Wypij D, McGowan FX Jr. The relationship between inflammatory activation and clinical outcome after infant cardiopulmonary bypass. Anesth Analg. 2010 Nov;111(5):1244-51. doi: 10.1213/ANE.0b013e3181f333aa. Epub 2010 Sep 9. PMID 20829561
- [Background] Bellomo R, Auriemma S, Fabbri A, D'Onofrio A, Katz N, McCullough PA, Ricci Z, Shaw A, Ronco C. The pathophysiology of cardiac surgery-associated acute kidney injury (CSA-AKI). Int J Artif Organs. 2008 Feb;31(2):166-78. doi: 10.1177/039139880803100210. PMID 18311733
- [Background] Blomquist S, Gustafsson V, Manolopoulos T, Pierre L. Clinical experience with a novel endotoxin adsorbtion device in patients undergoing cardiac surgery. Perfusion. 2009 Jan;24(1):13-7. doi: 10.1177/0267659109106730. PMID 19567543
- [Background] Peng ZY, Wang HZ, Carter MJ, Dileo MV, Bishop JV, Zhou FH, Wen XY, Rimmele T, Singbartl K, Federspiel WJ, Clermont G, Kellum JA. Acute removal of common sepsis mediators does not explain the effects of extracorporeal blood purification in experimental sepsis. Kidney Int. 2012 Feb;81(4):363-9. doi: 10.1038/ki.2011.320. Epub 2011 Sep 14. PMID 21918497